CLINICAL TRIAL: NCT01076556
Title: A Phase I Feasibility Trial of Cyclophosphamide, Alvocidib (Flavopiridol) and Rituximab (CAR) in Patients With High Risk B-cell CLL/SLL
Brief Title: Cyclophosphamide, Alvocidib, and Rituximab in Treating Patients With High Risk B-Cell Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01373; NCI-2011-01373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 09089; CDR0000666448; OSU-09089; OSU 09089 (Other: Ohio State University Comprehensive Cancer Center); 8267 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage I Small Lymphocytic Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Small Lymphocytic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — cytokine inducible SH2-containing protein; alvocidib; Cyclophosphamide; Rituximab

ARMS (1):
- Treatment (rituximab, cyclophosphamide, alvocidib) (Experimental): Patients receive rituximab IV over 4 hours on days 1 (days 1-3 in course 1), cyclophosphamide IV over 30-60 minutes on days 1-3, and alvocidib IV over 4.5 hours on days 1 and 8 (day 8 only in course 1).
  Interventions: Drug: Alvocidib Hydrochloride; Drug: Cyclophosphamide; Other: Diagnostic Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Rituximab

INTERVENTIONS:
Drug: Alvocidib Hydrochloride — Given IV
  Other Names: 4H-1-Benzopyran-4-one, 2-(2-chlorophenyl)-5, 7-dihydroxy-8-(3-hydroxy-1-methyl-4-piperidinyl)-, hydrochloride, (-)-cis-; Flavopiridol Hydrochloride; HL-275; HMR 1275; L-86-8275; L-868275; MDL 107,826A; MDL-107826A
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83

SUMMARY:
This phase I trial is studying the side effects and the best dose of alvocidib when given together with cyclophosphamide and rituximab in treating patients with high risk B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Alvocidib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can also block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Other find cancer cells and help kill them or carry cancer-killing substances to them. Giving cyclophosphamide, alvocidib, and rituximab together may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicity and maximum-tolerated dose of treatment with cyclophosphamide, alvocidib, and rituximab in patients with high-risk B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma.

II. To determine the feasibility of administering this regimen as an outpatient regimen in these patients.

SECONDARY OBJECTIVES:

I. To determine the complete response rate, partial response rate, and minimal-residual disease-negative response rate in patients treated with this regimen.

II. To determine the pharmacokinetics of alvocidib and dexamethasone as part of this regimen.

III. To determine the immunologic effects of this regimen as measured by serial T-cell and NK-cell number, T-cell function, and immunoglobulin levels.

OUTLINE: This is a dose-escalation study of alvocidib.

Patients receive rituximab IV over 4 hours on days 1 (days 1-3 in course 1), cyclophosphamide IV over 30-60 minutes on days 1-3, and alvocidib IV over 4.5 hours on days 1 and 8 (day 8 only in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Blood samples are collected periodically for pharmacokinetic and pharmacodynamic studies.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic lymphocytic leukemia (CLL) or B-cell prolymphocytic leukemia* (PLL) arising from CLL

  * Patients must have documented B-cell lymphocytosis > 5 x 10^9/L at some point since initial diagnosis of CLL
  * Patients must have B-cells that co-express CD5 with CD19 or CD20
  * Patients who do not have dim sIg or CD23 expression on their leukemia cells should be examined for cyclin D1 over-expression or t(11;14) to rule out mantle cell lymphoma
* To be considered high risk, patients must meet the following criteria:

  * At least 1 of the following:

    * 17p deletion
    * 11q deletion
    * Un-mutated IgV_H (≥ 98% homology)
    * Age > 70 years
    * B_2M > 4
  * AND at least 1 of the following:

    * Progressive or marked splenomegaly and/or lymphadenopathy
    * Anemia (hemoglobin < 11 g/dL) or thrombocytopenia (platelets < 100,000/mm^3)
    * Weight loss exceeding 10% of body weight over preceding 6 months
    * NCI grade 2 or 3 fatigue
    * Fevers > 100.5° F or night sweats for > 2 weeks without evidence of infection
    * Progressive lymphocytosis, with an increase exceeding 50% over a 2-month period or a doubling time of < 6 months
* No other concurrent hormones, chemotherapy, or radiotherapy except for steroids for new adrenal failure or hormones for nondisease-related conditions (e.g., insulin for diabetes)

  * No requirement for chronic corticosteroids
* ECOG performance status 0-2
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.5 times normal unless due to Gilbert disease, hemolysis, or disease infiltration of the liver
* AST ≤ 2 times normal unless due to hemolysis or disease infiltration of the liver
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No secondary or other malignancy that will limit survival to < 2 years
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No uncompensated HIV without adequate CD4 (> 200/mm^3) and requiring HIV medication
* No active hepatitis B infection
* No known G6PD deficiency
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to alvocidib, cyclophosphamide, rituximab, or other agents used in this study
* No prior alvocidib
* No prior purine analog therapy
* No more than 1 prior treatment with a biologic or alkylating agent
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of combination therapy with Cyclophosphamide, Alvocidib, and Rituximab | 21 days
  Determined using the CTEP Active Version of the CTCAE.
Treatment related adverse events assessed using the CTEP Active Version of the CTCAE | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Flynn, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States